CLINICAL TRIAL: NCT06722391
Title: Neuromuscular Electrical Stimulation: A Novel Treatment for Improving Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Principal Investigator, Sudip Bajpeyi, Professor, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2205558
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Insulin Resistance
Keywords: Neuromuscular Electrical Stimulation; Glucose Continuous Monitor; Blood Glucose; Obesity; Resting Metabolic rate
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Control (Placebo Comparator): Participants will receive stimulation only up to sensory level.
  Interventions: Device: Neuromuscular Electrical Stimulation (Sensory)
- NMES (Experimental): Participants will receive stimulation up to maximum tolerable level.
  Interventions: Device: Neuromuscular Electrical Stimulation
- Resistance Training (Placebo Comparator): Participants will receive exercise training with stimulation up to sensory level.
  Interventions: Device: Neuromuscular Electrical Stimulation (Sensory); Other: Resistance Training
- Resistance Training + NMES (Experimental): Participants will receive exercise training with stimulation up to maximum tolerable intensity.
  Interventions: Device: Neuromuscular Electrical Stimulation; Other: Resistance Training

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation (Sensory) — Group will receive Electrical Stimulation up to sensory level
  Other Names: Control
  Arms: Control; Resistance Training
Device: Neuromuscular Electrical Stimulation — Group will receive Electrical Stimulation up to maximum tolerable level
  Other Names: NMES Group
  Arms: NMES; Resistance Training + NMES
Other: Resistance Training — Group will receive exercise training.
  Other Names: Control
  Arms: Resistance Training; Resistance Training + NMES

SUMMARY:
Once written consent is obtained, the participant will be provided with an accelerometer to be worn for 7 days to assess current physical activity levels. Subjects will be provided with a standardized diet (55/15/30% CHO/PRO/FAT) prior to collection of pre-intervention data of insulin sensitivity. Individuals will then participate in an 8-week electrical stimulation intervention (30min/day, 3x/week) and randomized into placebo/control, NMES, resistance training combined with NMES (RT +NMES), or resistance training (RT) group (n=20 per group), followed by collection of post-intervention data. The control group will receive electrical stimulation up to sensory level, the NMES group will receive stimulation up to tolerable intensity to induce visible muscle contraction, the RT+ NMES will receive stimulation up to tolerable intensity during resistance training, and the RT group will only receive exercise training. Control and NMES group will self administer stimulation at home. Pre-and post-intervention data includes measurements for body composition, resting metabolic rate, VO2max, insulin sensitivity, and comprehensive blood work.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/Obese (BMI ≥25)
* Sedentary Lifestyle: Physical Activity Level<1.4
* Less than 150min/week of structured Exercise

Exclusion Criteria:

* Use of anti-hypertensive, lipid-lowering or insulin sensitizing medications
* Excessive alcohol, drug abuse, smoking
* Pregnant Women
* Unwilling to adhere to the study Intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | 8 weeks
  Insulin Sensitivity will be measured through repeated blood sampling during an Oral Glucose Tolerance Test and Continuous Glucose Monitoring

SECONDARY OUTCOMES:
Respiratory Exchange Ratio | 8 Weeks
  Respiratory Exchange Ratio will be used to quantify substrate utilization (fats vs carbohydrates) through the use of indirect calorimetry of in vivo gas exchange
Amount of lean mass | 8 weeks
  Amount of lean mass will be measured by dual energy x-ray absortiometry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No